CLINICAL TRIAL: NCT02389816
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase III Study to Evaluate the Efficacy and Safety of Once Daily Oral Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: A Phase 3 Study of Lu AA21004 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004/CCT-004; U1111-1167-1520 (Registry Identifier: WHO); JapicCTI-152831 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Major Depressive Disorder
Keywords: Drug therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo tablets, orally, once daily for up to Week 8
  Interventions: Drug: Placebo
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg tablets, orally, once daily for up to Week 8
  Interventions: Drug: Vortioxetine
- Vortioxetine 20 mg (Experimental): Vortioxetine 10 mg tablets, orally, once daily for up to Week 1 followed by vortioxetine 20 mg tablets, orally, once daily for up to Week 8
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Placebo — Placebo tablets
  Arms: Placebo
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: Lu AA21004
  Arms: Vortioxetine 10 mg; Vortioxetine 20 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of two fixed doses of vortioxetine (Lu AA21004; 10 or 20 mg/day) after 8 weeks of treatment in patients with major depressive disorder (MDD) in Japan.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, phase III study to assess the efficacy and safety of 8-week treatment of two fixed doses of Vortioxetine (Lu AA21004; 10 or 20 mg/day) in Japanese participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant suffers from recurrent MDD as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.3x).
4. The participant is a man or a woman aged 20 to 75 years (both inclusive) at the time of informed consent.
5. The reported duration of the current major depressive episode is 3 to 12 months (both inclusive) at the start of screening period.
6. The participant has a MADRS total score ≥26, Hamilton Depression Rating Scale (HAM-D17) total score ≥18, and Clinical global impression scale-Severity (CGI-S) score ≥4 at the start of screening period, at the start of placebo lead-in period and at the start of double-blind treatment period.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent to the end of the follow-up period.

Exclusion Criteria:

1. The participant has any following current or past history of psychiatric disorder and/or neurological disorder:

   * Any current psychiatric disorder other than MDD as defined by DSM-IV-TR (To be assessed by Mini International Neuropsychiatric Interview: MINI). A participant who exhibits symptoms of anxiety is eligible unless the participant fulfills the diagnostic criteria for a current anxiety disorder per DSM-IV-TR.
   * Current diagnosis or history of manic, mixed or hypomanic episode, MDD with psychotic features, schizophrenia or any other psychotic disorder (including substance-related mental disorders, or mental disorders due to a general medical condition) as defined by DSM-IV-TR.
   * Current diagnosis or history of any substance-related disorder (except nicotine and caffeine-related disorders) as defined by DSM-IV-TR.
   * The participant with a positive urine drug screening result at the start of screening period or the start of placebo lead-in period. In case that a participant showed positive test result at the start of screening period because the test was conducted before washout of pretreatment drug, the participant is eligible as long as he/she shows negative result at the start of placebo lead-in period.
   * Presence or history of any clinically significant neurological disorder (including epilepsy).
   * Any neurodegenerative disorder (e.g. Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease).
   * Any DSM-IV-TR axis II disorder.
2. The participant has the current or previous major depressive episode which was considered by the investigator or sub-investigator to have been resistant to 2 or more adequate antidepressants treatments of at least 6 weeks duration each at sufficient doses.
3. The participant has received any augmentation therapy (e.g. lithium, T3/T4, lamotrigine, sodium valproate, carbamazepine, additional atypical antipsychotic, or concomitant use of other antidepressant, etc.) for the current major depressive episode.
4. In the opinion of the investigator or sub-investigator, the participant has experienced significant number of major depressive episodes in the past, and is suspected of disease other than MDD.
5. In the opinion of the investigator or sub-investigator, the participant has experienced the first major depressive episode at his/her young age, and is suspected of disease other than MDD.
6. The participant has a MADRS total score at the start of double-blind treatment period that has improved or aggravated by 25% or more from the score at the start of placebo lead-in period.
7. The participant is significantly non-compliant with the study drug in the placebo lead-in period; e.g., not taking the study drug for 6 or more consecutive days.
8. The participant has received electroconvulsive therapy, vagus nerve stimulation, or repetitive transcranial magnetic stimulation therapy within 6 months prior to the screening period, or plans to initiate such therapy during the study.
9. The participant is receiving cognitive-behavioral therapy or psychotherapy at the time of informed consent, or plans to initiate such therapy during the study.
10. The participant is at significant risk of suicide or has a score ≥5 on Item 10 (suicidal thoughts) of the MADRS at the start of screening period, at the start of placebo lead-in period or at the start of double-blind treatment period, or has attempted suicide within 6 months prior to the start of screening period.
11. The participant has experienced any environmental change (e.g. temporary retirement, returnment, change of residence) considered by the investigator or sub-investigator to have the potential to impact on the efficacy evaluation, or plans such environmental changes during the study.
12. The participant is currently receiving drug therapy for thyroid dysfunction.
13. The participant is currently receiving hormonal therapy for gynecological disease.
14. The participant has taken excluded medications during the protocol-specified period, or will require to take excluded medications during the study.
15. The participant has previously received vortioxetine.
16. The participant has received study drug in a previous clinical study of Lu AA21004 (including this study).
17. The participant has a clinically significant chronic liver disease.
18. The participant has a history of severe allergy or hypersensitivity to drugs.
19. The participant has a clinically significant unstable illness, for example, liver disorder or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, neoplastic, skin and subcutaneous tissue disorders, eye disorders, or metabolic disturbance.
20. The participant has clinically significant abnormal vital signs as determined by the investigator or sub-investigator at the start of screening period, placebo lead-in period, or double-blind treatment period.
21. The participant has clinically significant abnormal electrocardiogram (ECG) as determined by the investigator or sub-investigator, at the start of the screening period, at the start of placebo lead-in period, or at the start of double-blind treatment period.
22. The participant has clinically significant abnormal findings of clinical laboratory tests as determined by the investigator or sub-investigator, or has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × ULN at the start of screening period or at the start of placebo lead-in period.
23. If female, the participant is pregnant or lactating.
24. The participant has a disease or takes medications that could, in the opinion of the investigator or sub-investigator, interfere with the evaluation of the safety, tolerability, or efficacy.
25. The participant is, in the opinion of the investigator or sub-investigator, unsuitable for this study for any other reason.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (47):
- Japan (47):
  - Nagoya, Aichi-ken
  - Nagareyama, Chiba
  - Noda, Chiba
  - Iizuka, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Kōriyama, Fukushima
  - Shirakawa, Fukushima
  - Sapporo, Hokkaido
  - Ashiya, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Kurashiki, Okayama-ken
  - Kadoma, Osaka
  - Kita-ku, Osaka
  - Sakai, Osaka
  - Sayama, Osaka
  - Karatsu, Saga-ken
  - Kawagoe, Saitama
  - Kusatsu, Shiga
  - Anan, Tokushima
  - Arakawa-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Hachiōji, Tokyo
  - Itabashi-ku, Tokyo
  - Katsushika-ku, Tokyo
  - Koto-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Mitaka, Tokyo
  - Musashino, Tokyo
  - Nakano-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Suginami-ku, Tokyo
  - Taito-ku, Tokyo
  - Toshima-ku, Tokyo
  - Kofu, Yamanashi
  - Fukuoka
  - Hiroshima
  - Kumamoto
  - Okayama
  - Saitama

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Watanabe K, Fujimoto S, Marumoto T, Kitagawa T, Ishida K, Nakajima T, Moriguchi Y, Fujikawa K, Inoue T. Therapeutic Potential of Vortioxetine for Anhedonia-Like Symptoms in Depression: A Post Hoc Analysis of Data from a Clinical Trial Conducted in Japan. Neuropsychiatr Dis Treat. 2022 Feb 19;18:363-373. doi: 10.2147/NDT.S340281. eCollection 2022. PMID 35221687
- [Derived] Inoue T, Fujimoto S, Marumoto T, Kitagawa T, Ishida K, Nakajima T, Moriguchi Y, Fujikawa K, Watanabe K. Therapeutic Potential of Vortioxetine for Anxious Depression: A Post Hoc Analysis of Data from a Clinical Trial Conducted in Japan. Neuropsychiatr Dis Treat. 2021 Dec 21;17:3781-3790. doi: 10.2147/NDT.S335028. eCollection 2021. PMID 34992372
- [Derived] Inoue T, Fujimoto S, Marumoto T, Kitagawa T, Ishida K, Nakajima T, Moriguchi Y, Fujikawa K, Watanabe K. Early Improvement with Vortioxetine Predicts Response and Remission: A Post Hoc Analysis of Data from a Clinical Trial Conducted in Japan. Neuropsychiatr Dis Treat. 2021 Dec 18;17:3735-3741. doi: 10.2147/NDT.S340309. eCollection 2021. PMID 34955641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 64 investigative sites in Japan, from 10 April 2015 to 16 March 2018.
Pre-assignment Details: Participants with a historical diagnosis of major depressive disorder were enrolled placebo lead-in period for one week prior to randomization, after that participants randomized and enrolled in one of three treatment group (Placebo Group, vortioxetine 10 milligrams (mg) Group, vortioxetine 20 mg Group) for 8 weeks as double-blind treatment period.
Groups:
- Vortioxetine 20 mg: Vortioxetine 10 mg tablets, orally, once daily for up to Week 1, followed by vortioxetine 20 mg tablets, orally, once daily for up to Week 8
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Started | 164 | 165 | 164
Completed | 149 | 152 | 152
Not Completed | 15 | 13 | 12
Not completed — Randomized but Not Treated | 1 | 0 | 0
Not completed — Pretreatment Event or Adverse Event (AE) | 4 | 6 | 7
Not completed — Major Protocol Deviation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal of Consent | 6 | 4 | 4
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Non Compliance with Study Drug | 1 | 1 | 1
Not completed — Reason not Specified | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set, Randomized set was defined as all participants who randomized in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg | Total
Number analyzed (Participants) | 164 | 165 | 164 | 493
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (10.47) | 40.0 (10.58) | 40.4 (11.31) | 40.0 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 72 | 80 | 224
  Male | 92 | 93 | 84 | 269
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 164 | 165 | 164 | 493
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 166.5 (8.51) | 165.2 (9.04) | 164.5 (7.86) | 165.4 (8.51)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 62.44 (12.218) | 61.97 (12.958) | 61.54 (12.006) | 61.98 (12.382)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 22.44 (3.450) | 22.56 (3.560) | 22.65 (3.594) | 22.55 (3.530)
Montgomery Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension). MADRS corresponds to core symptoms of depression, and rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 30.5 (3.87) | 30.8 (3.73) | 30.6 (3.62) | 30.6 (3.73)
Hamilton Depression Scale (HAM-D17) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The HAM-D17 is a clinician-rated scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 where a higher score indicates a greater depressive state. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 22.0 (3.19) | 22.1 (3.10) | 22.2 (3.10) | 22.1 (3.13)
Clinical Global Impressions-Severity (CGI-S) Score [Mean (Standard Deviation); unit: Scores on a scale] — The CGI-S assesses the impression of the participant's current state of mental illness. The current severity of mental illness is rated on a seven-point scale (1=normal, not ill at all ~ 7=most extremely ill) based on a total clinical experience. Higher scores indicate greater severity of mental illness. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 4.5 (0.63) | 4.5 (0.63) | 4.5 (0.61) | 4.5 (0.62)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: Scores on a scale] — The SDS assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 13.9 (6.22) | 14.0 (6.00) | 14.8 (5.47) | 14.2 (5.91)
Digit Symbol Substitution Test (DSST) Score [Mean (Standard Deviation); unit: Scores on a scale] — The DSST is a neuropsychological test to assess cognitive function. Participants are required to copy symbols that are paired with simple geometric shapes or numbers within a specific time for a total possible score of 0 to 133. Higher scores-correct number of symbols reflects greater objective cognitive functioning. An increase in score represents an improvement in an integrated measure of cognitive function. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 163 | 164 | 490
    (all) | 60.2 (13.93) | 56.8 (15.15) | 58.0 (13.72) | 58.3 (14.32)
Perceived Deficits Questionnaire (PDQ-5) Score [Mean (Standard Deviation); unit: Scores on a scale] — PDQ-5 is a self-administered 5-item questionnaire to assess cognition function, including subscales of attention/concentration, retrospective memory, prospective memory, and planning/organization. PDQ-5 total score ranges from 0 to 20 with smaller scores indicate greater cognitive function. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 163 | 165 | 164 | 492
    (all) | 9.0 (3.54) | 9.5 (3.52) | 9.7 (3.47) | 9.4 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score to Week 8
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension). MADRS corresponds to core symptoms of depression, and rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: Full Analysis Set (FAS): All participants who were randomized and received at least 1 dose of the study drug in the double-blind treatment period.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | -12.37 (0.714) | -15.03 (0.699) | -15.45 (0.705)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0080, Mixed Models Analysis; Mixed Models for Repeated Measures (MMRM); Least square (LS) mean difference = -2.66, 95% CI 2-sided [-4.63 to -0.70], Standard Error of Mean 0.999
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0023, Mixed Models Analysis; Mixed Models for Repeated Measures (MMRM); LS mean difference = -3.07, 95% CI 2-sided [-5.05 to -1.10], Standard Error of Mean 1.003

2. Secondary Outcome: MADRS Response at Week 8 (Last Observation Carried Forward (LOCF))
Description: Reported data was percentage of participants who met MADRS response criteria (defined as a ≥50% decrease in the MADRS total score from Baseline) at Week 8 for each group. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension). MADRS corresponds to core symptoms of depression, and rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Week 8
Population: FAS: All participants who were randomized and received at least 1 dose of the study drug in the double-blind treatment period. Here, number analyzed is the number of participants who were evaluable at each category.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Percentage of Participants | 36.6 | 47.9 | 50.6
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0341, Regression, Logistic; Odds Ratio (OR) = 1.621, 95% CI 2-sided [1.037 to 2.533]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0110, Regression, Logistic; Odds Ratio (OR) = 1.788, 95% CI [1.143 to 2.799]

3. Secondary Outcome: MADRS Remission at Week 8 (LOCF)
Description: Reported data was percentage of participants who met MADRS remission criteria (defined as a MADRS total score ≤10) at Week 8 for each group. MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension). MADRS corresponds to core symptoms of depression, and rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates improvement.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Percentage of Participants | 21.1 | 32.1 | 30.9
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0186, Regression, Logistic; Odds Ratio (OR) = 1.839, 95% CI 2-sided [1.107 to 3.054]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0418, Regression, Logistic; Odds Ratio (OR) = 1.700, 95% CI 2-sided [1.020 to 2.834]

4. Secondary Outcome: Change From Baseline in Hamilton Depression Scale (HAM-D17) Total Score to Week 8 (LOCF)
Description: The HAM-D17 is a clinician-rated scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 where a higher score indicates a greater depressive state.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | -8.38 (0.541) | -10.19 (0.524) | -10.17 (0.532)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0165, ANCOVA; LS mean difference = -1.81, 95% CI 2-sided [-3.290 to -0.332], Standard Error of Mean 0.753
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0190, ANCOVA; LS mean difference = -1.79, 95% CI 2-sided [-3.278 to -0.295], Standard Error of Mean 0.759

5. Secondary Outcome: Clinical Global Impressions-Improvement (CGI-I) Score at Week 8 (LOCF)
Description: The CGI-I assesses the participant's state of mental illness improvement. The participant's condition compared to baseline is rated on a seven-point scale (1=very much improved ~ 7=very much worse). Higher scores indicate greater worsening of illness. Values closest to 1 for this outcome measure indicate the greatest improvement of symptoms.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | 2.77 (0.085) | 2.42 (0.084) | 2.38 (0.085)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0031, ANCOVA; LS mean difference = -0.36, 95% CI 2-sided [-0.590 to -0.121], Standard Error of Mean 0.120
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0011, ANCOVA; LS mean difference = -0.39, 95% CI 2-sided [-0.629 to -0.158], Standard Error of Mean 0.120

6. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score to Week 8 (LOCF)
Description: The CGI-S assesses the impression of the participant's current state of mental illness. The current severity of mental illness is rated on a seven-point scale (1=normal, not ill at all ~ 7=most extremely ill) based on a total clinical experience. Higher scores indicate greater severity of mental illness.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | -1.19 (0.0088) | -1.42 (0.0087) | -1.48 (0.0087)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0609, ANCOVA; LS mean difference = -0.23, 95% CI 2-sided [-0.474 to 0.011], Standard Error of Mean 0.123
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0179, ANCOVA; LS mean difference = -0.29, 95% CI 2-sided [-0.537 to -0.051], Standard Error of Mean 0.124

7. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score to Week 8 (LOCF)
Description: The SDS assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | -2.85 (0.447) | -4.20 (0.432) | -4.43 (0.440)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0311, ANCOVA; LS mean difference = -1.34, 95% CI 2-sided [-2.564 to -0.122], Standard Error of Mean 0.621
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0126, ANCOVA; LS mean difference = -1.57, 95% CI 2-sided [-2.807 to -0.339], Standard Error of Mean 0.628

8. Secondary Outcome: Change From Baseline in Digit Symbol Substitution Test (DSST) Total Score to Week 8 (LOCF)
Description: The DSST is a neuropsychological test to assess cognitive function. Participants are required to copy symbols that are paired with simple geometric shapes or numbers within a specific time for a total possible score of 0 to 133. Higher scores-correct number of symbols reflects greater objective cognitive functioning. An increase in score represents an improvement in an integrated measure of cognitive function.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | 4.92 (0.632) | 4.13 (0.628) | 4.80 (0.629)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.3793, ANCOVA; LS mean difference = -0.79, 95% CI 2-sided [-2.539 to 0.968], Standard Error of Mean 0.893
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.9011, ANCOVA; LS mean difference = -0.11, 95% CI 2-sided [-1.862 to 1.641], Standard Error of Mean 0.891

9. Secondary Outcome: Change From Baseline in Perceived Deficits Questionnaire (PDQ-5) Total Score to Week 8 (LOCF)
Description: PDQ-5 is a self-administered 5-item questionnaire to assess cognition function, including subscales of attention/concentration, retrospective memory, prospective memory, and planning/organization. PDQ-5 total score ranges from 0 to 20 with smaller scores indicate greater cognitive function.
Time Frame: Baseline (At the start of double-blind treatment period), up to 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 164 | 165 | 164
Scores on a scale | -1.41 (0.234) | -2.28 (0.231) | -2.69 (0.234)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority; p = 0.0089, ANCOVA; LS mean difference = -0.87, 95% CI 2-sided [-1.512 to -0.218], Standard Error of Mean 0.329
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority; p = 0.0001, ANCOVA; LS mean difference = -1.27, 95% CI 2-sided [-1.922 to -0.619], Standard Error of Mean 0.332

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/165 | 2/163
Serious Adverse Events (participants affected / at risk) | 1/161 | 1/165 | 3/163
Other Adverse Events (participants affected / at risk) | 32/161 | 54/165 | 51/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Vortioxetine 10 mg (N=165) | Vortioxetine 20 mg (N=163)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=161) | Vortioxetine 10 mg (N=165) | Vortioxetine 20 mg (N=163)
Nausea (Gastrointestinal disorders) | 1 | 21 | 25
Vomiting (Gastrointestinal disorders) | 0 | 9 | 6
Nasopharyngitis (Infections and infestations) | 26 | 23 | 21
Somnolence (Nervous system disorders) | 6 | 7 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT02389816/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02389816/SAP_001.pdf